CLINICAL TRIAL: NCT02302469
Title: A Multicenter Phase I/II Dose Escalation Study of Lenalidomide in Relapse/Refractory Waldenstrom Macroglobulinemia
Brief Title: Study of Lenalidomide in Relapse/Refractory Waldenstrom Macroglobulinemia
Acronym: RV-WM-0426
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008_15/0837; 2008-006370-15 (EudraCT Number)
Record Dates: First submitted 2014-06-24; First posted 2014-11-27 (Estimated); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Waldenstrom Macroglobulinemia
Keywords: Lenalidomide; Hematology; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- revlimid (Other): a dose-escalation of revlimid
  Interventions: Drug: Revlimid

INTERVENTIONS:
Drug: Revlimid — Three cohorts of subjects will be successively exposed to escalating doses of Lenalidomide (15, 20 and 25mg once daily on days 1-21 of a 28 day cycle).
  Other Names: lénalidomide

SUMMARY:
The purpose of this study is to determine the recommended dose of lenalidomide in subjects with relapse and refractory Waldenstrom Macroglobulinemia.

DETAILED DESCRIPTION:
Waldenstrom Macroglobulinemia (lymphoplasmacytic lymphoma, WM) is a low-grade lymphoplasmacytic lymphoma characterized by the involvement of the bone marrow with lymphoplasmacytic cells and the production of immunoglobulin M monoclonal protein in the circulation . Waldenstrom Macroglobulinemia is characterized by anemia and cytopenias due in part to the clonal expansion in the bone marrow. In addition, infiltration of the liver, spleen, and lymph nodes may occur in 15-20% of the patients leading to enlargement of these organs. Finally, complications related to elevated serum monoclonal protein such as hyperviscosity may also occur. Waldenstrom macroglobulinemia is an incurable disease with an overall median survival of 5-6 years from the development of symptoms . The median age at diagnosis is 63 years Options of therapy in patients with relapsed/refractory Waldenstrom Macroglobulinemia include rituximab, alkylating agents, nucleoside analogues. Although novel agents, such as bortezomib and thalidomide, are still matter of debate, several phase II studies have demonstrated that novel agents, especially Bortezomib, are active agent in relapsed and refractory Waldenstrom Macroglobulinemia .The overall response rate in single agents bortezomib studies reach 80%, with major responses observed in 30-40% of patients. Therefore, there is a need to identify new therapeutic agents for Waldenstrom Macroglobulinemia patients.

In view of their success in the treatment of patients with Multiple Myeloma, immunomodulatory drugs (IMiDS) were tested in patients with Waldenstrom Macroglobulinemia, although their experience is limited. Thalidomide is nonmyelosuppressive, immunomodulatory, and antiangiogenic and may be a reasonable choice for patients for whom first-line therapies have failed, those who have had disease relapse and are not candidates for alkylating or nucleoside analogue therapy, or patients with pancytopenia . Twenty three Waldenstrom Macroglobulinemia patients were evaluable in a phase II study of thalidomide in combination with rituximab. Although the overall and major response rates were of 78% and 70%, respectively; tolerance was a concern, and dose reduction of thalidomide occurred in all patients and led to discontinuation in 11 patients.

Lenalidomide has been studied in Multiple Myeloma and myelodysplastic syndrome and found to be more potent and also to lack the neurotoxic and prothrombotic adverse effects of thalidomide . Based on the potent activity of lenalidomide in Multiple Myeloma and the lack of neuropathy with this agent, and based on the interesting results reported with thalidomide-rituximab phase II tril in relapse/refractory Waldenstrom Macroglobulinemia, a phase II study of lenalidomide 25mg daily in combination with rituximab was perform in patients with relapsed/refractory Waldenstrom Macroglobulinemia. Lenalidomide was administered for 3 weeks, followed by a one week pause for an intended duration of 48 weeks. Patients received one week of therapy with lenalidomide, after which rituximab (375mg/m2) was administered weekly on weeks 2-5, then 13-16 . Twelve patients were evaluable for an overall and a major response rate of 67% and 33%, and a median time to progression of 15.6 months. Acute decreases in hematocrit were observed during first 2 weeks of lenalidomide therapy in 13/16 (81%) patients with a median hematocrit decrease of 4.4% (1.7-7.2%). Despite reduction of initiation doses to 5mg daily, anemia continued to be problematic without evidence of hemolysis or more general myelosuppression. Therefore, the mechanism for pronounced anemia in Waldenstrom Macroglobulinemia patients receiving lenalidomide remains to be determined and the use of this agent among Waldenstrom Macroglobulinemia patients remains investigational.

ELIGIBILITY:
Inclusion Criteria:

The most important criteria for patient eligibility include:

1. Age >=18 years
2. Patients must have received prior therapy (any number of therapies) for WM and have relapsed or refractory WM
3. Eastern Cooperative Oncology Group performance score of 0 - 2
4. Hemoglobin >= 10g/dL or hematocrit >= 30%
5. Absolute neutrophil count (ANC) >1000/mm3 and platelet count >75,000/mm3
6. Adequate organ function defined as

   * serum glutamate pyruvate transaminase and serum glutamate oxaloacetate transaminase < 2 x International Unit/l
   * Total bilirubin >= 1.5 mg/dL
   * Clearance creatinin > 50 ml/mn
7. Evaluable immunochemical abnormalities including abnormal electrophoresis and serum free light chain assay with an increase of either kappa or lambda light chain lev -

Exclusion Criteria:

Key Exclusion criteria

1. Any other uncontrolled medical condition or comorbidity that might interfere with subject's participation
2. Patients treated or requiring corticosteroids >30mg/day
3. Pregnant or breast feeding females (Lactating females must agree not to breast feed while taking lenalidomide)
4. Use of any other experimental drug or therapy within 28 days of baseline
5. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
6. Known positive for HIV or infectious hepatitis, type A, B or C -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants with dose limiting toxicities (DLT) of lenalidomide as a Measure of Safety and Tolerability. | 1 month
  To determine the recommended dose of lenalidomide in subjects with relapse and refractory Waldenstrom Macroglobulinemia

SECONDARY OUTCOMES:
number of patients with a response to lenalidomide | 60 months
  Response rate will be evaluated following standard criteria for evaluation of response in Waldenstrom Macroglobulinemia recommended by the Second International Waldenstrom Macroglobulinemia Workshop will be used in this study
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 60 months
  Safety (type, frequency, severity, and relationship of adverse events to study treatment). Incidence of Treatment Emergent Adverse Event (TEAE), Serious Adverse Event (SAE) and laboratory abnormalities
Measurements of free light chain assays. | Baseline, 2 months, 3 months
  To explore the value of frequent measurements of free light chain assays at baseline and after the first 2 cycles, then every 3 cycles and its relationship to response rate.
Response duration. | 60 months
  • Response duration (time between first documentation of response and disease progression). Time to disease progression (from the date of the first dose to the date of the first observation of disease progression).
progression free survival | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: TOURNILLAC Olivier, Dr, Principal Investigator — Centre Hospitalier CLERMOND FERRAND; MOREL Pierre, Dr, Principal Investigator — Centre Hospitalier de Lens; LELEU Xavier, Dr, Study Director — CHRU LILLE; LEGOUILL Steven, Dr, Principal Investigator — Centre Hospitalier de NANTES; LEBLOND Véronique, Dr, Principal Investigator — APHP PARIS; BANOS Anne, Dr, Principal Investigator — Centre Hospitalier de BAYONNE; SALLES Gilles, Pr, Principal Investigator — Centre Hospitalier de LYON
Locations (7):
- France (7):
  - Centre Hospitalier de la côte basque, Bayonne
  - Ch Clermond Ferrand, Clermont-Ferrand
  - CH LENS, Lens
  - Chru Lille, Lille
  - Ch Nantes, Nantes
  - Groupe hospitalier Pitié Salpétrière, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fouquet G, Guidez S, Petillon MO, Louni C, Ohyba B, Dib M, Poulain S, Herbaux C, Martin A, Thielemans B, Brice P, Choquet S, Bakala J, Bories C, Demarquette H, Nudel M, Tournilhac O, Arnulf B, LeGouill S, Morel P, Banos A, Karlin L, Salles G, Leblond V, Leleu X. Lenalidomide is safe and active in Waldenstrom macroglobulinemia. Am J Hematol. 2015 Nov;90(11):1055-9. doi: 10.1002/ajh.24175. Epub 2015 Oct 6. PMID 26284823
- See also: European Clinical Trials Register — https://www.clinicaltrialsregister.eu/ctr-search/search?query=CHRU++RV+WM